CLINICAL TRIAL: NCT04571723
Title: Health Mindset as a Driver of Efficacy of a Diabetes Prevention Program in the Blackfeet Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-13
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: One group will receive the original diabetes prevention program curriculum, and other group will receive modified health mindset curriculum.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blind to the condition they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Established Diabetes Prevention Program (Active Comparator): This arm will receive the established diabetes prevention program curriculum.
  Interventions: Behavioral: Diabetes Prevention Program
- Health Mindset modified Diabetes Prevention Program (Active Comparator): This arm will receive the modified curriculum with the added health mindset information.
  Interventions: Behavioral: Health Mindset modified diabetes prevention program

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — This is the established Diabetes prevention program curriculum.
  Arms: Established Diabetes Prevention Program
Behavioral: Health Mindset modified diabetes prevention program — This is the established diabetes prevention program curriculum with the addition of curriculum focused on the role of mindset in health.
  Arms: Health Mindset modified Diabetes Prevention Program

SUMMARY:
The overall goal of this project is to understand whether the established Diabetes prevention program works to reduce diabetes risk by shifting mindsets about health.

DETAILED DESCRIPTION:
The Diabetes Prevention Program (DPP), a lifestyle intervention which aims to modify health behaviors, has reduced diabetes risk across several American Indian Communities. However, there were significant attrition rates, and non-completers were at the highest risk at baseline. One's mindset about health (i.e. whether it is fixed or malleable) may affect their likelihood of completing the intervention and its efficacy in reducing risk. With an existing CAB, I will develop a culturally congruent adaptation of the DPP, the Mindset-DPP (M-DPP). The M-DPP will include a discussion of mindset in each session and will present material focused on the plasticity of health, including evidence that one's mindset can affect outcomes that relate to risk for diabetes. The investigators will implement the DPP and the MDPP in a sample of 40 Blackfeet community members at risk for diabetes and test whether the M-DPP associates with greater shifts towards a growth health mindsets (i.e. health can be changed by effort) compared to the DPP, and whether the M-DPP associates with greater increases in physical activity levels and greater reductions in waist circumference, and greater retention compared to the standard DPP.

ELIGIBILITY:
Inclusion Criteria:

* self identified as American Indian
* identified as high risk for diabetes based on the American Diabetes Association paper and pencil test
* must reside on the Blackfeet reservation

Exclusion Criteria:

-chronic disease diagnosis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Health Mindset | baseline, 6 weeks after baseline, and immediately after the intervention (11 weeks after baseline)
  The Health Mindset Questionnaire will be used to measure the degree to which participants view health as fixed or modifiable. Higher scores on the scale reflect a stronger growth health mindset (i.e. health can be changed) while lower numbers reflect a more fixed health mindset (i.e. health is not modifiable). The range of possible scores is 3-18. Change will be calculated from subtracting the health mindset score will be calculated by subtracting the health mindset score at baseline from subsequent health mindset scores (2 change scores will be calculated: one at 6 weeks after baseline and one at 11 weeks after baseline).

SECONDARY OUTCOMES:
physical activity levels | during the intervention, up to 11 weeks.
  accelerometer derived measure of average physical activity levels
waist circumference | baseline, 6 weeks after baseline, and immediately after the intervention (11 weeks after baseline)
  circumference of the waist will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Blackfeet Community College, Browning, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided